CLINICAL TRIAL: NCT06805864
Title: Pembrolizumab Concurrent With and Following Carbon-ion Radiotherapy for Locally Advanced Cervical Adenocarcinoma (BROTHER STUDY)
Brief Title: Pembrolizumab Concurrent With and Following Carbon-ion Radiotherapy for Locally Advanced Cervical Adenocarcinoma
Acronym: BROTHER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gunma University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Tatsuya Ohno, Professor, Department of Radiation Oncology, Gunma University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2024-049
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma
Keywords: Cervical Cancer; Carbon-ion Radiotherapy; Pembrolizumab
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CIRT＋CDDP＋Pembro (Experimental): Patients will first be treated with 16 fractions/4 weeks of carbon-ion radiation therapy (CIRT) followed by 3 cycles/2 weeks of image-guided brachytherapy (IGBT). During this radiation therapy, up to 5 cycles of weekly cisplatin will be given concurrently.
  In addition to these, pembrolizumab will be administered every 3 weeks at 200 mg for the first 2 cycles, then increased to 400 mg every 6 weeks for 17 cycles over 2 years.
  Interventions: Drug: Pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Drug: Pembrolizumab (KEYTRUDA®) — Pembrolizumab is administered at 200 mg every 3 weeks for the first 2 cycles during Chemo-CIRT, after completion of radiotherapy, the dose is increased to 400 mg and given every 6 weeks for a total of 17 cycles over 2 years.

SUMMARY:
The goal of this clinical trial is to learn if pembrolizumab works for cervical adenocarcinoma treat with concurrent chemo-carbon-ion radiaotherapy (CIRT).

The main questions it aims to answer are:

• Does concurrent chemo-CIRT with pembrolizumab improves 2-year progression-free survival (PFS), compared with concurrent chemoradiotherapy with conventional X-rays?

ELIGIBILITY:
Inclusion Criteria:

* 1. Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed adenocarcinoma or adenosquamous carcinoma of the uterine cervix and Stage ⅡA2, ⅡB, ⅢA, ⅢB, ⅢC1r, IVA according to FIGO classification (2018) will be enrolled in this study.

  2. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.

  3. Have measurable disease based on RECIST 1.1.

  4. Archival tumor tissue sample or a newly obtained biopsy of a tumor lesion that was not previously irradiated was provided. Formalin-fixed, paraffin-embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsy samples are preferred to archived tissues.

  5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of pembrolizumab.

  6. Have adequate organ function below. Specimens must be collected within 10 days to the start of pembrolizumab administration.
* Absolute neutrophil count (ANC) ≥ 1500/µL, Platelets ≥ 100000/µ, Hemoglobin ≥9.0 g/dL or ≥ 5.6 mmol/L, Creatinine clearance ≥ 50 mL/min, Total bilirubin ≤1.5 ×ULN or direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN, AST and ALT ≤2.5 × ULN, International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.

Exclusion Criteria:

* 1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).

  2. Has received prior radical surgery, RT, or systemic therapy (including investigational drugs) for cervical cancer. Note: Conization for localized cervical tumors is allowed.

  3. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.

Note: please refer to Section 5.3 for information on COVID-19 vaccines

4. Has received an investigational agent or has used an investigational device within 4 weeks prior to pembrolizumab administration.

5. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab.

6. Known additional malignancy that is progressing or has required active treatment within the past 3 years.

Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.

7. Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.

8. Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (e.g.., thyroxine, insulin, or physiologic corticosteroid).

9. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.

10. Has an active infection requiring systemic therapy.

11. History of active Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as detectable HCV RNA [qualitative]) infection.

12. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.

13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

14. Is pregnant or breast feeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

15. Has had an allogenic tissue/solid organ transplant.

16. History of HIV infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | At 2 years after the start of trial treatment
  It is based on the investigator's RECIST 1.1 assessment, or in the absence of imaging evidence of disease progression based on RECIST 1.1, histologically confirmed PD, after concurrent chemo-CIRT with pembrolizumab.

SECONDARY OUTCOMES:
Overall survival (OS) | At 2 years after the start of trial treatment
  To evaluate the 2-year overall survival after concurrent chemo-CIRT with pembrolizumab.
Complete response (CR) rate | At 6 months after the start of trial treatment
  To evaluate the complete response (CR) rate, defined as the maximum response of the primary tumor based on RECIST 1.1 assessment at 6 months after initiation of CIRT.
Local control (LC) | At 2 years after the start of trial treatment
  To evaluate the 2-year local control (LC) after concurrent chemo-CIRT with pembrolizumab.
Acute and late toxicities | Acute (≤ 90 days) and late toxicities (> 90 days) over 2 years after the start of trial treatment.
  To evaluate the acute and late toxicities of concurrent chemo-CIRT with pembrolizumab.

CONTACTS AND LOCATIONS:
Locations (1):
- Gunma University Hospital, Maebashi, Gunma, Japan

IPD SHARING:
Plan to Share IPD: No